CLINICAL TRIAL: NCT01472809
Title: A Randomized, Double Blind Placebo Controlled Phase 1 Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of ZYGK1, a Novel Glucokinase Activator, Following Oral Administration in Healthy Volunteers
Brief Title: A Clinical Study to Evaluate Safety, Tolerability and Pharmacokinetics of Oral ZYGK1 in Healthy Volunteers
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Not achieved the objective till 4 mg single dose
Sponsor: Zydus Lifesciences Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZYGK1/1001; CTRI/2011/12/002249 (Other: Clinical Trial Registry India)
Record Dates: First submitted 2011-11-09; First posted 2011-11-17 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Diabetes
Keywords: ZYGK1; Cadila; Zydus; ZRC; Zydus Research Center; Phase 1; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo
- ZYGK1 (Experimental): ZYGK1 tablets; 0.125, 0.25, 0.5, 1, 2, ... mg.
  Dose escalation will continue till single AE occurs in any block of 3 volunteers on ZYGK1 or pharmacokinetic (dose linearity) saturation is reached or desired PK/PD effect is achieved
  Interventions: Drug: ZYGK1

INTERVENTIONS:
Drug: ZYGK1 — ZYGK1 Tablets: 0.125, 0.25, 0.5, 1, 2, .... mg.
  Dose escalation will continue till single AE occurs in any block of 3 volunteers on ZYGK1 or pharmacokinetic (dose linearity) saturation is reached or desired PK/PD effect is achieved
  Arms: ZYGK1
Drug: Placebo — Placebo Tablets: 0.125, 0.25, 0.5, 1, 2, ... mg
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine (1) whether ZYGK1 is safe and well tolerated, (2) the pharmacokinetics (what body does to ZYGK1) and (3) pharmacodynamics (what drugs does to the body) in the healthy and diabetic subject.

DETAILED DESCRIPTION:
This study will be a randomized, double blind, placebo controlled study and is divided into four plans:

1. Plan I: Single Ascending Dose (SAD) Study
2. Plan II: Multiple Ascending Dose (MAD)Study
3. Plan III: Gender Effect study
4. Plan IV: Food Effect study

First Plan I, Plan III and Plan IV will be conducted in healthy volunteers. After reviewing the results, decision shall be taken whether the multiple ascending doses shall be studied in healthy human volunteers or in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-45 years
2. Mentally, physically, and legally eligible to give informed consent
3. Male and female volunteers weighing between 50-75 kg and 45-75 kg (4) respectively.
4. Ability to communicate effectively with the study personnel
5. Willingness to adhere to the protocol requirements
6. For gender effect study, only females with history of sterility or at least one year menopause or use of long acting nonhormonal contraceptive measures (e.g., intrauterine device) will be recruited.
7. At least one panel, in single ascending dose and multiple ascending dose will include subjects with type 2 diabetes as defined by American Diabetes Association

Exclusion Criteria:

1. Presence or history of hypersensitivity to any of the active or inactive ingredients of ZYGK1 formulation
2. Presence or history of pancreatitis at any time (Serum Amylase/Serum Lipase more than upper normal limit (UNL))
3. Presence or history of severe gastrointestinal disease in the last 6 months
4. Presence or history of renal insufficiency at any time (serum creatinine >UNL)
5. Active liver disease and/or liver transaminases greater than 1.5 X UNL
6. History or presence of other systemic disorders or diseases (e.g., respiratory, gastrointestinal, endocrine, immunological, dermatological, neurological, psychiatric disease or any other body system involvement)
7. Abnormal bleeding time (BT), clotting time (CT), prothrombin time (PT), and activated partial prothrombin time (APTT)
8. History or presence of any medication in the last 14 days
9. History or presence of significant alcoholism or drug abuse within the past 1 year
10. History or presence of significant smoking (more than 10 cigarettes per day) or consumption of tobacco products (more than 10 times per day)
11. Difficulty with donating blood
12. Systolic blood pressure more than 140 mmHg and less than 100 mmHg and diastolic blood pressure more than 90 mmHg and less than 60 mmHg
13. Pulse rate less than 60 minute and more than 100/minute
14. Any clinically significant laboratory findings during screening
15. History or presence of any clinically significant electrocardiogram (ECG) abnormalities during screening
16. Major illness and/or major surgery in last 3 months
17. Volunteers who have participated in any drug research study other than the present trial within past 3 months
18. Volunteers who have donated one unit (350 ml) of blood in the past 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Upto 14 Days
  Safety and tolerability for-
  * Plan I, Plan III and Plan IV [Time frame: up to Day 8]
  * Plan II [Time frame: upto Day 14]
  Frequency of adverse events will be assessed at each dose level.

SECONDARY OUTCOMES:
Pharmacokinetics | 7 Days
  Pharmacokinetics after oral administration of ZYGK1 in
  * Plan I, III and IV: [Time frame: 0.25 - 168 hrs post drug administration]
  * Plan II: [Time frame:Day 1: 0.25 - 12 hours, Day 2-6: 0, 2, 4 Hours, Day: 0.25-168 hours post drug administration]
  Effects of food on the pharmacokinetics will be assessed in healthy subjects.
Pharmacodynamics | 7 Days
  Plasma glucose, serum insulin, C-peptide and glucagoan estimate -
  * Plane I and Plan III [Time frame: Day 0 and Day 1: upto 4 hours post oral glucose 75 grams]
  * Plan II [Time frame: Day 0, Day 1 and Day 7: upto 4 hours post oral glucose 75 grams]
  * Plan IV: [Time frame: Period 2: Day 0 and Day 1: upto 4 hours post meal]

CONTACTS AND LOCATIONS:
Overall Officials: Rajendrakumar H Jani, PhD(Medical), Study Director — Clinical R&D, Zydus Research Center, Cadila Healthcare Limited, Moraiya, Ahmedabad-382213, Gujarat, India; Kevinkumar Kansagra, MD, Principal Investigator — Clinical R&D, Zydus Research Center, Cadila Healthcare Limited, Moraiya, Ahmedabad-382213, Gujarat, India
Locations (1):
- Clinical R&D, Zydus Research Center, Cadila Healthcare Limited, NH No.8, Moraiya, Ahmedabad, Gujarat, India